CLINICAL TRIAL: NCT00856323
Title: Biobehavioral Interventions for HIV-negative Methamphetamine-using MSM
Brief Title: Contingency Management for Methamphetamine Abstinence and HIV Post-Exposure Prophylaxis in Men Who Have Sex With Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 702632
Record Dates: First submitted 2009-03-03; First posted 2009-03-05 (Estimated); Results first posted 2012-11-27 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-08

CONDITIONS: Amphetamine-Related Disorders; HIV; HIV Infections
Keywords: Methamphetamine; HIV; Post-exposure prophylaxis; HIV seronegativity
MeSH Terms: conditions — Amphetamine-Related Disorders; HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEP/CM (Experimental): Participants are provided contingency management vouchers for methamphetamine abstinence, and can initiate postexposure prophylaxis (Truvada; 1 pill daily for 28 days) after non-occupational exposure to HIV.
  Interventions: Drug: Truvada; Behavioral: CM

INTERVENTIONS:
Drug: Truvada — At qualifying exposure, participants will take 28 days' worth (at one pill per day) of 200 mg emtricitabine and 300 mg tenofovir DF (Truvada).
  Other Names: Emtricitabine and tenofovir disoproxil fumarate
Behavioral: CM — Participants will submit a urine sample every Monday, Wednesday, and Friday for 8 weeks (a total of 24 urine samples). Samples will be tested for methamphetamine metabolites.
  Other Names: Contingency Management

SUMMARY:
This study seeks to decrease methamphetamine use and concomitant high-risk sexual behaviors among methamphetamine-using men who have sex with men (MSM) by combining a biomedical intervention with a behavioral intervention. The behavioral intervention will consist of an 8-week course of contingency management (CM) through which participants will be reinforced for testing negative for methamphetamine metabolites during periodic urine analyses. The biomedical intervention involves a 28-day course of an antiretroviral drug (Truvada) to be administered after an unanticipated HIV risk exposure (i.e., engaging in either receptive or insertive anal sex without a condom with someone who is HIV-positive or of unknown status). In combining these two interventions, this study seeks to evaluate the combined intervention's effects on sexual risk behaviors and methamphetamine use.

DETAILED DESCRIPTION:
At the baseline, all eligible participants underwent informed consent; completed baseline assessments; received rapid HIV testing; provided specimens for syphilis, gonorrhea and chlamydia testing; and received a medical examination. Those who reported a high-risk sexual or drug exposure episode with an HIV-positive or serostatus-unknown source within the preceding 72 hours immediately initiated postexposure prophylaxis. All other participants received a 4-day ''starter pack'' of Truvada to be initiated only in the case of a future high-risk exposure to HIV. All participants began the voucher-based CM intervention upon study entry. For the initial 8 weeks of study conduct, participants presented to the study site three times weekly for a urine drug screen for methamphetamine metabolites. Participants who provided urine samples that were negative for methamphetamine metabolites earned vouchers, which escalated in value for successive negative urine samples. A participant with a missing sample or a sample positive for methamphetamine metabolites did not earn vouchers. Accrued vouchers were never forfeited and could be redeemed at any time during the study for gift certificates or goods or services that promote healthy, pro-social behaviors; vouchers could not be redeemed for cash.

ELIGIBILITY:
Inclusion Criteria:

* Individual must identify as a male who has sex with other men (MSM);
* At least 18 years of age;
* HIV negative serostatus on baseline rapid oral HIV antibody test;
* Self-reported methamphetamine use within the previous 72 hours and test positive for methamphetamine metabolites at baseline;
* Self-reported unprotected anal intercourse (either receptive or insertive) with an HIV-positive or status unknown partner within the previous 3 months;
* Self-reports no previous hypersensitivity to any of the components of Truvada (tenofovir disoproxil fumarate or emtricitabine);
* Willing to comply with study requirements (i.e., monitored urine testing three times per week, meet with physician within first week of enrollment, begin medication immediately following an unexpected high-risk sexual exposure, and contact the clinic and meet with physician within 92 hours of unexpected high-risk sexual exposure).

Exclusion Criteria:

* Does not identify as a male who has sex with other men;
* Under 18 years of age;
* HIV positive, by self-report or as indicated by the results on the baseline rapid oral HIV antibody test;
* Self-reports any previous hypersensitivity to any of the components of Truvada;
* Has not used methamphetamine in the previous 72 hours and does not test positive for methamphetamine metabolites;
* Has not had unprotected anal intercourse with an HIV-positive or status unknown partner within the previous 3 months;
* Unwilling to comply with study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy J Reback, Ph.D., Principal Investigator — Friends Research Institute, Inc.; Raphael J Landovitz, M.D., Principal Investigator — UCLA Center for Clinical AIDS Research and Education; Steve Shoptaw, Ph.D., Principal Investigator — UCLA Department of Family Medicine
Locations (1):
- Friends Community Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Landovitz RJ, Fletcher JB, Inzhakova G, Lake JE, Shoptaw S, Reback CJ. A novel combination HIV prevention strategy: post-exposure prophylaxis with contingency management for substance abuse treatment among methamphetamine-using men who have sex with men. AIDS Patient Care STDS. 2012 Jun;26(6):320-8. doi: 10.1089/apc.2011.0432. PMID 22680280
- [Derived] Fletcher JB, Rusow JA, Le H, Landovitz RJ, Reback CJ. High-risk Sexual Behavior is Associated with Post-Exposure Prophylaxis Non-adherence among Men who have Sex with Men Enrolled in a Combination Prevention Intervention. J Sex Transm Dis. 2013;2013:210403. doi: 10.1155/2013/210403. PMID 24527254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2009 and August 2010, 358 individuals inquired about the study on the basis of recruitment efforts, 64 presented for screening, and 53 participants enrolled in the study.
Pre-assignment Details: Reasons for Screen Failure (N = 7): HIV-positive at baseline screening; negative urine screen for methamphetamine§; did not complete baseline assessments; provided incorrect information at phone screening.
Groups:
- PEP/CM: Truvada : At qualifying exposure, participants will take 28 days' worth (at one pill per day) of 200 mg emtricitabine and 300 mg tenofovir DF (Truvada).
  CM : Participants will submit a urine sample every Monday, Wednesday, and Friday for 8 weeks (a total of 24 urine samples). Samples will be tested for methamphetamine metabolites.
Period: Overall Study
Arm/Group | PEP/CM
Started | 53
Completed | 51
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | PEP/CM
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 53
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 53
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Methamphetamine Use in Previous 30 Days.
Description: Mean number of days (of the past 30) of methamphetamine use.
Time Frame: 3-months after baseline
Population: 53 enrolled and 2 were withdrawn.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PEP/CM
Number analyzed (Participants) | 51
days | 1.6 (2.4)

2. Secondary Outcome: Description of Incident STI Infections.
Description: Proportional 3-month incidence of syphilis, rectal gonorrhea, pharyngeal gonorrhea, and rectal Chlamydia.
Time Frame: Baseline and 3-months
Population: 53 enrolled and 2 were withdrawn.
Measure: Mean (Full Range); unit: Proportion of Participants
Arm/Group | PEP/CM
Number analyzed (Participants) | 51
Proportion of Participants | .074 [.045 to .114]

3. Secondary Outcome: HIV-related Sexual Risk Behaviors in Previous 30 Days.
Description: Self-reported episodes of Unprotected Anal Intercourse in the previous 30 days.
Time Frame: 3-months after baseline
Population: 53 enrolled and 2 were withdrawn.
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | PEP/CM
Number analyzed (Participants) | 51
episodes | .44 (1.4)

4. Secondary Outcome: Post-Exposure Prophylaxis Medication Adherence
Description: Median medication adherence rate, defined as the proportion of pills taken relative to the number of pills prescribed (i.e., # of pills taken / # of pills prescribed).
Time Frame: 28-days
Population: 35 participants initiated PEP
Measure: Median (Inter-Quartile Range); unit: proportional medication adherence
Arm/Group | PEP/CM
Number analyzed (Participants) | 35
proportional medication adherence | 0.96 [0.57 to 1.0]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | PEP/CM
Serious Adverse Events (participants affected / at risk) | 2/53
Other Adverse Events (participants affected / at risk) | 4/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEP/CM (N=53)
depression (Psychiatric disorders) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEP/CM (N=53)
abdominal pain (Gastrointestinal disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 1 (1)
flatulence (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No